CLINICAL TRIAL: NCT01454843
Title: A Prospective Eye to Eye Comparison of LASIK Using the Alcon Allegretto Wavefront-Guided Excimer Laser Versus AMO Visx Wavefront-Guided Excimer Laser
Brief Title: LASIK Using the Alcon Allegretto Wavefront-Guided Excimer Laser vs AMO Visx Wavefront-Guided Excimer Laser
Acronym: LASIK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Edward E. Manche, Professor of Ophthalmology, Stanford University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21220
Record Dates: First submitted 2011-10-06; First posted 2011-10-19 (Estimated); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Myopia; Astigmatism
Keywords: Myopia; Astigmatism; Aberrations; Wavefront; LASIK; Wavefront LASIK
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wavefront-guided LASIK - Allegretto (Active Comparator): Wavefront-guided LASIK using the Allegretto excimer laser.
  Interventions: Procedure: Wavefront-guided LASIK - Allegretto
- Wavefront-guided LASIK - AMO (Active Comparator): Wavefront-guided LASIK using AMO CustomVue excimer laser.
  Interventions: Procedure: Wavefront-guided LASIK - AMO

INTERVENTIONS:
Procedure: Wavefront-guided LASIK - Allegretto — Wavefront-guided LASIK using the Allegretto excimer laser for myopia.
  Other Names: Alcon Wavelight Allegretto Eye-Q 400 Hz excimer laser
  Arms: Wavefront-guided LASIK - Allegretto
Procedure: Wavefront-guided LASIK - AMO — Wavefront-guided LASIK using the AMO CustomVue excimer laser for myopia.
  Other Names: AMO Visx CustomVue S4 IR excimer laser
  Arms: Wavefront-guided LASIK - AMO

SUMMARY:
The purpose of the study is to compare the results of LASIK surgery when using Alcon Allegretto wavefront-guided excimer laser system compared to AMO Visx Custom wavefront-guided excimer laser system in patients with nearsightedness with and without astigmatism.

DETAILED DESCRIPTION:
The patients will have a comprehensive eye examination once they express an interest in the study. This includes a slit lamp examination of the front of the eye and a dilated fundoscopic examination of the back of the eye. if there is any pathology noted that would exclude the patient from the study, then we will inform the patient and make an appropriate referral. If the patient is deemed appropriate for the study after a comprehensive examination included computerized videokeratography, then they can be enrolled. The patient will undergo bilateral simultaneous eye surgery. Which eye is treated with a wavefront-guided excimer laser and which eye is treated with wavefront-optimized will be randomized so there is a 50% chance for either eye to receive one treatment. The patients will be seen on the day of surgery, post op day one, post op day 4-7, one month, three months, six months and one year. The patient will receive topical antibiotics in each eye for one week following the procedure. LASIK treated eyes will receive pred forte 1% ophthalmic drops for one week after treatment. All of this is within the usual and customary standard of care for the treatment of patients undergoing lasik surgery.

The research procedures are the least risky that can be performed consistent with sound research design.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 21 and older with healthy eyes.
* Nearsightedness between -0.50 diopters and -7.00 diopters with or without astigmatism of up to 3.50 diopters.

Exclusion Criteria:

* Subjects under the age of 21.
* Patients with excessively thin corneas.
* Patients with topographic evidence of keratoconus.
* Patients with ectatic eye disorders.
* Patients with autoimmune diseases.
* Patients who are pregnant or nursing.
* Patients must have similar levels of nearsightedness with or without astigmatism in each eye.
* They can not be more than 1.5 diopters of difference between eyes.
* Patients must have similar levels of astigmatism in each eye.
* They can not have more than 1.5 diopters of difference in nearsightedness or astigmatism between their two eyes.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-04-01 (Actual); Primary Completion 2011-03-31 (Actual); Study Completion 2012-06-23 (Actual)

PRIMARY OUTCOMES:
Efficacy | 1 year
  Efficacy measures uncorrected visual acuity following the LASIK surgery. We will record how many eyes see 20/40, 20/30, 20/25, 20/20, 20/16, 20/12.5 and 20/10 after the surgery without glasses or contact lenses. We are measuring how well patients see after the surgery without glasses or contact lenses.

SECONDARY OUTCOMES:
Low contrast visual acuity | 1 year
  Measuring changes in best spectacle corrected low contrast visual acuity (5 and 25 percent).
Higher order aberrations | 1 year
  Measure changes in higher order aberrations.
Safety | One year
  Will will assess safety by measuring change in best spectacle corrected visual acuity. We will record the number of eyes that gain, lose or have no change in the best spectacle corrected visual acuity after the surgery. This is measured using snellen visual acuity charts. The ideal outcome would be that there were no loss of any lines of best spectacle corrected visual acuity and a high percentage of gains of lines of best spectacle corrected visual acuity.
Predictability | One year
  Percentage of eyes within +/- 0.5 diopters of the intended correction

CONTACTS AND LOCATIONS:
Overall Officials: Edward E Manche, MD, Principal Investigator — Stanford University
Locations (1):
- Byers Eye Institute at Stanford, Palo Alto, California, United States

REFERENCES:
- [Background] He L, Manche EE. Contralateral eye-to-eye comparison of wavefront-guided and wavefront-optimized photorefractive keratectomy: a randomized clinical trial. JAMA Ophthalmol. 2015 Jan;133(1):51-9. doi: 10.1001/jamaophthalmol.2014.3876. PMID 25321951
- [Background] He L, Manche EE. Prospective randomized contralateral eye evaluation of subjective quality of vision after wavefront-guided or wavefront- optimized photorefractive keratectomy. J Refract Surg. 2014 Jan;30(1):6-12. doi: 10.3928/1081597X-20131217-01. PMID 24868564
- [Background] Lee WS, Manche EE. Comparison of simulated keratometric changes following wavefront-guided and wavefront-optimized myopic laser-assisted in situ keratomileusis. Clin Ophthalmol. 2018 Mar 29;12:613-619. doi: 10.2147/OPTH.S161387. eCollection 2018. PMID 29636597
- [Background] He L, Liu A, Manche EE. Wavefront-guided versus wavefront-optimized laser in situ keratomileusis for patients with myopia: a prospective randomized contralateral eye study. Am J Ophthalmol. 2014 Jun;157(6):1170-1178.e1. doi: 10.1016/j.ajo.2014.02.037. Epub 2014 Feb 19. PMID 24560995
- [Background] Sales CS, Manche EE. One-year outcomes from a prospective, randomized, eye-to-eye comparison of wavefront-guided and wavefront-optimized LASIK in myopes. Ophthalmology. 2013 Dec;120(12):2396-2402. doi: 10.1016/j.ophtha.2013.05.010. Epub 2013 Jun 15. PMID 23778091
- [Background] Sales CS, Manche EE. One-year eye-to-eye comparison of wavefront-guided versus wavefront-optimized laser in situ keratomileusis in hyperopes. Clin Ophthalmol. 2014 Nov 12;8:2229-38. doi: 10.2147/OPTH.S70145. eCollection 2014. PMID 25419115